

## educAR

Validation of a strategy to improve therapeutic adherence in rheumatoid arthritis.

Informed consent form

Version: v2 27/12/2021

## INFORMED CONSENT FORM

## EDUCAR PROJECT: VALIDATION OF A STRATEGY TO IMPROVE THERAPEUTIC ADHERENCE IN RHEUMATOID ARTHRITIS Me ..... ..... (name and patient's last name). I have read the information sheet given to me. I was able to ask questions about the study. I have received enough information about the study. I have spoken with I understand that my participation is voluntary. I understand that I can withdraw from the study: 1. - Whenever I want. 2. - Without having to explain. 3. - Without this affecting my medical care. I freely give my consent to participate in the study. **PATIENT:**

| SignatureDate |
|----------------------------------------|
| Name and surname (IN CAPITAL LETTERS) |
| ······································ |
| RESEARCHER: |
| SignatureDate |
| Name and surname (IN CAPITAL LETTERS) |

| WITNESS: |
|------------------------------------------------------------------|
| Signature |
| Name and surname (IN CAPITAL LETTERS) |
| SECTION FOR THE REVOCATION OF CONSENT |
| Me, |
| I revoke the consent to participate in the process, signed above |